CLINICAL TRIAL: NCT05905718
Title: Comparison of the Immediate Effects of Spinomed Orthosis and Biofeedback Orthosis on Balance and Walking Performance in Elderly Individuals With Thoracic Hyperkyphosis
Brief Title: The Effects of Spinomed Orthosis and Biofeedback Orthosis in Elderly Individuals With Thoracic Hyperkyphosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Kader Eldemir, Doctor Physiotherapist, Ordu University
Other Study IDs: Spinomed-Biofeedback orthosis
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Elderly People
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinomed orthosis group
  Interventions: Other: assessment
- Biofeedback orthosis group
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment — Assessments of thoracic kyphosis angle, balance performance, and gait performance.

SUMMARY:
Hyperkyphosis, defined as excessive sagittal curvature of the thoracic spine, is the most common spinal deformity in elderly individuals. The prevalence of hyperkyphosis in elderly individuals is reported to be between 20% and 40%. Hyperkyphosis affects the mobility, walking, and balance of the individual negatively and causes changes in the physical performance of elderly individuals. Therefore, it is important to evaluate and treat hyperkyphosis in elderly people. One of the approaches to treating people with hyperkyphosis is the use of spinal orthoses such as the Spinomed orthosis and Biofeedback orthosis. Regular use of spinal orthoses reduces the angle of kyphosis by 11%. In addition, spinal orthoses help increase walking speed and distance, improve balance, and prevent falls. Spinomed and Biofeedback soft posture orthoses are spinal orthoses used in the treatment of kyphotic posture. Studies on Spinomed orthosis have demonstrated that it strengthens postural muscles, and therefore also prevents falls. Soft orthoses, which provide feedback, provide a warning to the individual through sound or vibration when the spinal alignment of the individual is disturbed, and provide the correction of posture with active muscle strength. However, little evidence exists regarding the effect of these two orthoses on improving balance and walking performance in elderly people with thoracic hyperkyphosis. Therefore, this study was developed to enable a comparison of the effect of the Spinomed orthosis and the biofeedback orthosis on balance and walking performance in elderly people with thoracic hyperkyphosis.

DETAILED DESCRIPTION:
Volunteer healthy elderly individuals between the ages of 60-80 will be recruited into our study and the individuals will be randomly divided into two groups Spinomed orthosis and postural orthosis which provides biofeedback. In both groups, balance and gait assessments with or without orthosis will be done twice.

ELIGIBILITY:
Inclusion Criteria:

* having an age of 60 years or above
* the ability to walk at least 10 meters independently
* thoracic hyperkyphosis angle above 40 degrees
* Mini-mental test score greater than 24

Exclusion Criteria:

* having fractures or surgery on the spine or lower limbs within the last 12 months
* having degenerative impairment in the spine, such as scoliosis and osteoarthritis
* having any neurological and cognitive impairment

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly people with thoracic hyperkyphosis will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2023-09-09 (Actual)

PRIMARY OUTCOMES:
Balance assessment without the orthosis | at baseline
  The Balance Performance Tests, which are performed using computerized posturography, measure postural sway and limit of stability in response to static and dynamic conditions, are measured using a force platform.
Balance assessment with the orthosis | 1.5 hours after applying orthosis
  The Balance Performance Tests, which are performed using computerized posturography, measure postural sway and limit of stability in response to static and dynamic conditions, are measured using a force platform.
Gait assessment without the orthosis | at baseline
  Gait parameters will be assessed via the G-Walk on two separate occasions. The G-Walk is a device that is worn on the waist via an elastic belt. The G-Walk has with a triaxial accelerometer,, a triaxial magnetometer, and a triaxial gyroscope. This hardware is capable of acquiring and transmitting data to a computer through a Bluetooth connection and at the end of each analysis an automatic report containing the gait assessment results is ready to be analyzed.
Gait assessment with the orthosis | 1.5 hours after applying orthosis
  Gait parameters will be assessed via the G-Walk on two separate occasions. The G-Walk is a device that is worn on the waist via an elastic belt. The G-Walk has with a triaxial accelerometer,, a triaxial magnetometer, and a triaxial gyroscope. This hardware is capable of acquiring and transmitting data to a computer through a Bluetooth connection and at the end of each analysis an automatic report containing the gait assessment results is ready to be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No